CLINICAL TRIAL: NCT05805423
Title: ENDOblock: Do Bilateral Superficial Cervical Blocks With Local Wound Infiltration Decrease Postoperative Pain After Thyroid Surgery
Brief Title: ENDOblock: Bilateral Superficial Cervical Blocks With Local Wound Infiltration in Thyroid Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1958184
Record Dates: First submitted 2023-03-14; First posted 2023-04-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Post Operative Pain; Nausea and Vomiting, Postoperative; Opioid Use
Keywords: bilateral superficial cervical plexus block; post operative pain after thyroidectomy
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Intervention Model Description: single center, prospective, double-blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bilateral superficial cervical plexus blocks + local wound infiltration (Experimental): the bilateral superficial cervical plexus block will be performed with 10mL of 0.25% Bupivacaine injected bilaterally (total 20mL) at Erb's point in the lateral neck, which is located at the mid-point between the mastoid process and the posterior border of the clavicular head of the sternocleidomastoid muscle. The injection is just below the lateral border of the sternocleidomastoid muscle, which produces surface level anesthesia of the neck, targeting superficial nerves of the cervical plexus. Then 10mL of 0.25% Bupivacaine will be injected at the planned neck incision (local wound infiltration) on the anterior neck. These will be done intra-operative and only once
  Interventions: Procedure: bilateral superficial cervical plexus blocks and local wound infiltration
- placebo + local wound infiltration (Placebo Comparator): 10mL of 0.25% bupivacaine injected at the planned neck incision (local wound infiltration), with 10mL of normal saline injected at bilateral Erb's point (total 20mL) (placebo at site of BSCPB). These will be done intra-operative and only once.
  Interventions: Procedure: placebo injection and local wound infiltration

INTERVENTIONS:
Procedure: bilateral superficial cervical plexus blocks and local wound infiltration — 10mL bupivacaine at Erb's point bilaterally and 10mL 0.25% Bupicacaine at incision
  Arms: Bilateral superficial cervical plexus blocks + local wound infiltration
Procedure: placebo injection and local wound infiltration — 10mL normal saline at Erb's point bilaterally and 10mL 0.25% Bupicacaine at incision
  Arms: placebo + local wound infiltration

SUMMARY:
This is a single center, prospective, double-blinded randomized controlled trial comparing the efficacy of bilateral superficial cervical plexus blocks (BSCPB) with local wound infiltration vs placebo with local wound infiltration in reducing thyroid surgery postoperative pain. Primary outcomes assessed are post operative pain, quality of life/recovery, post operative nausea/vomiting and opioid use.

DETAILED DESCRIPTION:
The study consists of enrollment period until 74 participants acquired (37 will be in each arm), a treatment period (day of surgery), and a 2 week follow up period.

A web-based randomizer (https://randomizer.org/) will be used to randomly assign participants into Group A (bilateral superficial cervical plexus blocks + local wound infiltration) and Group B (placebo + local wound infiltration). Numbered envelopes with respective assignments and medications sealed within will be prepared by a research assistant separate from the surgical team and brought to the operating theater together with subjects. Participants and surgeons will both be blinded to the intervention.

Induction of anesthesia will occur prior to performing a block. All participants will be closely monitored by anesthesia, including BP, HR, SpO2, tidal volumes, peak pressures, CO2.

Participants who are randomized to the bilateral superficial cervical plexus blocks + local wound infiltration (Group A) will have 10mL of 0.25% Bupivacaine injected bilaterally (total 20mL) at Erb's point, which is located at the mid-point between the mastoid process and the posterior border of the clavicular head of the sternocleidomastoid muscle (SCM). The injection is just below the lateral border of the SCM, which produces surface level anesthesia of the neck, targeting superficial nerves of the cervical plexus (1). Injections will be aimed at just below the dermis. Then 10mL of 0.25% Bupivacaine will be injected at the planned neck incision (local wound infiltration). The participants randomized to the placebo+local wound infiltration group will have 10mL of 0.25% Bupivacaine injected at the planned neck incision, with 10mL of normal saline injected at bilateral Erb's point (total 20mL). All injections will be performed by the same team of two surgeons and with 22 gauge needles to standardize the technique. Surgery will be performed according to standard clinical care, also by the same group of surgeons, standardizing the surgical technique.

As is our standard practice following thyroid surgery, participants will be observed for at least 4 hours in the post anesthesia care unit for postoperative complications, adequate pain control, neck hematoma, and possible complications from the BSCPB. These rare complications can include CNS toxicity, partial brachial plexus palsy, Horner's syndrome, or recurrent laryngeal nerve block. All participants will be assessed at 3-5 hours after surgery to ensure their post operative pain is acceptable on oral medications and they do not have any of the above complications. They will either stay overnight or be discharged home with standardized discharge instructions and pain medication regimen, which will include taking Tylenol every 6 hours, alternated with ibuprofen. This pain regimen will be used for participants unless changed for clinical contraindications as determined by the attending surgeon. If participants request additional medication, they will be prescribed with a few pills of 5mg oxycodone, which they can take up to every 4 hours.

A primary outcome will be postoperative pain. Neck pain intensity will be quantified using the numeric rating scale (visual analog score 0-10, VAS) at 3-5 hours (in post anesthesia care unit), post operative day 2, via telephone call, and 2 weeks +/- 3 days postoperatively (at their follow up video visit). In addition, comparisons between groups will be made for 48-hour opioid usage by participants self-reporting at the post operative day 2 follow up phone call.

Another primary outcome is the 15-item quality of recovery questionnaire score at post operative day 2 and two weeks postoperative.

Incidence of nausea, vomiting, dysphagia or hoarseness in the first 2 days after surgery will also be measured (roughly the first 48 hours after surgery).

The planned data analysis for quality of recovery scores will be done using independent t test, with 95% confidence interval and two-tailed p values reported. Significance levels will be set at p=0.05. The investigators plan to analyze pain scores across the 3 periods with linear regression, with output the difference between the groups across all periods (95% CI and p=0.05) and the difference between the groups in each period (95% CI and p=0.05). The 48-hour opioid usage will be likely analyzed by using independent t test with 95% confidence intervals and two-tailed p values reported (p=0.05). Nausea, vomiting, hoarseness, dysphagia will be recorded as categorical variables and the investigators plan to analyze them using the Pearson chi-squared test.

ELIGIBILITY:
Inclusion Criteria:

* undergoing thyroid surgery, either hemi- or total thyroidectomy
* over 18 years-old and
* able to consent for themselves

Exclusion Criteria:

* have had previous neck surgery
* have coagulation disorders
* on anticoagulants
* are pregnant
* allergic to bupivacaine
* anyone with chronic pain conditions
* has received steroid injections or used opioids/pain medications in the two weeks leading up to surgery
* have a substernal goiters
* undergoing lateral neck lymph node dissection
* unable to take NSAIDs
* kidney dysfunction (defined as GFR <60) within 90 days of surgery, prohibiting the use of NSAIDs

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
does the addition of bilateral superficial cervical plexus blocks with local wound infiltration decrease postoperative pain after thyroid surgery | assessed at 3-5 hours (in post anesthesia care unit [PACU])
  Neck pain intensity will be quantified using the numeric rating scale (visual analog score 0-10, VAS). Higher scores mean more pain. Lower scores are a better outcome
does the addition of bilateral superficial cervical plexus blocks with local wound infiltration decrease postoperative pain after thyroid surgery | post operative day 2, via telephone call
  Neck pain intensity will be quantified using the numeric rating scale (visual analog score 0-10, VAS). Higher scores mean more pain. Lower scores are a better outcome
does the addition of bilateral superficial cervical plexus blocks with local wound infiltration decrease postoperative pain after thyroid surgery | 2 weeks +/- 3 days postoperatively (at their follow up video visit)
  Neck pain intensity will be quantified using the numeric rating scale (visual analog score 0-10, VAS). Higher scores mean more pain. Lower scores are a better outcome
does the addition of bilateral superficial cervical plexus blocks with local wound infiltration increase patient quality of life/recovery after thyroid surgery | post operative day 2, via telephone call
  15-item Quality of recovery (QoR) after anesthesia is a validated self reported measure of the early postoperative health status of patients. highest score possible 150, lowest 0. higher score means better quality of life and recovery
does the addition of bilateral superficial cervical plexus blocks with local wound infiltration increase patient quality of life/recovery after thyroid surgery | 2 weeks +/- 3 days postoperatively (at their follow up video visit)
  15-item Quality of recovery (QoR) after anesthesia is a validated self reported measure of the early postoperative health status of patients. highest score possible 150, lowest 0. higher score means better quality of life and recovery
Incidence of nausea and/or vomiting post operatively | assessed at 3-5 hours (in post anesthesia care unit [PACU])
  patients are given a questionnaire assessing level of nausea on scale 0-10, higher score is more nauseated and worse outcome. yes/no question if they have vomited since surgery and how many times. more episodes of vomiting is worse outcome.
Incidence of nausea and/or vomiting post operatively | post operative day 2 via telephone
  patients are given a questionnaire assessing level of nausea on scale 0-10, higher score is more nauseated and worse outcome. yes/no question if they have vomited since surgery and how many times. more episodes of vomiting is worse outcome.
Incidence of nausea and/or vomiting post operatively | 2 weeks +/- 3 days postoperatively (at their follow up video visit)
  patients are given a questionnaire assessing level of nausea on scale 0-10, higher score is more nauseated and worse outcome. yes/no question if they have vomited since surgery and how many times. more episodes of vomiting is worse outcome.

SECONDARY OUTCOMES:
hoarseness | assessed at 3-5 hours (in post anesthesia care unit [PACU])
  yes/no question on survey- yes answer is worse outcome
hoarseness | post operative day 2, via telephone call
  yes/no question on survey- yes answer is worse outcome
dysphagia (difficulty swallowing) | assessed at 3-5 hours (in post anesthesia care unit [PACU])
  yes/no question on survey- yes answer is worse outcome
dysphagia (difficulty swallowing) | post operative day 2, via telephone call
  yes/no question on survey- yes answer is worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JS, Ko JS, Bang S, Kim H, Lee SY. Cervical plexus block. Korean J Anesthesiol. 2018 Aug;71(4):274-288. doi: 10.4097/kja.d.18.00143. Epub 2018 Jul 4. PMID 29969890
- [Background] Mayhew D, Sahgal N, Khirwadkar R, Hunter JM, Banerjee A. Analgesic efficacy of bilateral superficial cervical plexus block for thyroid surgery: meta-analysis and systematic review. Br J Anaesth. 2018 Feb;120(2):241-251. doi: 10.1016/j.bja.2017.11.083. Epub 2017 Dec 5. PMID 29406173
- [Background] Dieudonne N, Gomola A, Bonnichon P, Ozier YM. Prevention of postoperative pain after thyroid surgery: a double-blind randomized study of bilateral superficial cervical plexus blocks. Anesth Analg. 2001 Jun;92(6):1538-42. doi: 10.1097/00000539-200106000-00038. PMID 11375842
- [Background] Karthikeyan VS, Sistla SC, Badhe AS, Mahalakshmy T, Rajkumar N, Ali SM, Gopalakrishnan S. Randomized controlled trial on the efficacy of bilateral superficial cervical plexus block in thyroidectomy. Pain Pract. 2013 Sep;13(7):539-46. doi: 10.1111/papr.12022. Epub 2012 Dec 19. PMID 23279371
- [Background] Cai HD, Lin CZ, Yu CX, Lin XZ. Bilateral superficial cervical plexus block reduces postoperative nausea and vomiting and early postoperative pain after thyroidectomy. J Int Med Res. 2012;40(4):1390-8. doi: 10.1177/147323001204000417. PMID 22971490
- [Background] Eti Z, Irmak P, Gulluoglu BM, Manukyan MN, Gogus FY. Does bilateral superficial cervical plexus block decrease analgesic requirement after thyroid surgery? Anesth Analg. 2006 Apr;102(4):1174-6. doi: 10.1213/01.ane.0000202383.51830.c4. PMID 16551919
- [Background] Myles PS, Shulman MA, Reilly J, Kasza J, Romero L. Measurement of quality of recovery after surgery using the 15-item quality of recovery scale: a systematic review and meta-analysis. Br J Anaesth. 2022 Jun;128(6):1029-1039. doi: 10.1016/j.bja.2022.03.009. Epub 2022 Apr 14. PMID 35430086